CLINICAL TRIAL: NCT00115102
Title: Sensory Examination and Pharmacological Modulation of Oral Hyperexcitability in Patients With Atypical Odontalgia and Matched Healthy Controls
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Pain Research Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: AO1
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Last update posted 2006-06-20 (Estimated); Status verified 2006-06

CONDITIONS: Odontalgia
Keywords: Atypical odontalgia; capsaicin; pain; neuropathic pain
MeSH Terms: conditions — Toothache; Pain; Neuralgia | interventions — Fentanyl; Esketamine

INTERVENTIONS:
Drug: fentanyl
Drug: S-ketamine

SUMMARY:
This project examines experimental pain and chronic pain in the mouth, specifically the condition called atypical odontalgia (AO:atypical toothpain). In 16 patients with AO and 16 healthy persons, capsaicin (chili-pepper) is applied to the gingiva to cause pain. This pain is evaluated by the participants. In three sessions, 3 different medications are tested for effect on the pain. The medications are fentanyl, S-ketamine and placebo-treatment (saline). The aim is to know more about pain mechanisms in AO in order to develop an effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Atypical odontalgia

Exclusion Criteria:

* BMI > 30
* Heart conditions
* Lung disease
* Diseases of the liver or kidneys
* Hypertension, untreated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-03; Study Completion 2005-10

PRIMARY OUTCOMES:
Pain
Sensitivity to heat and cold
Sensitivity to mechanical stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Troels Staehelin Jensen, MD, PhD, Dr.Sci, Study Chair — Aarhus University Hospital
Locations (1):
- Danish Pain Research Center, Aarhus, Denmark